CLINICAL TRIAL: NCT06678750
Title: Evaluation of Clinical Outcomes and Patient Recovery in Patients Receiving TKA With Traditional Instrumentation Systems Compared to Full Arc of Motion Gap Balancing Using the Newton™ Knee Protocol: A Prospective Clinical Study
Brief Title: A Prospective Clinical Study Evaluating the Newton™ TKA Protocol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding not finalized
Sponsor: Newton-Wellesley Hospital (Other)
Collaborators: Exactech (Industry)
Responsible Party: Principal Investigator, Christopher M. Melnic, MD, Principal Investigator, Newton-Wellesley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024p002323
Record Dates: First submitted 2024-10-30; First posted 2024-11-07 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2024-10

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Comparison Group: TKA patients whose surgery was conducted with traditional, manual instrumentation (Active Comparator): The comparison groups includes TKA patients whose surgery is conducted using traditional, manual, non-navigated instrumentation.
  Interventions: Procedure: TKA
- Intervention Group: Patients whose TKA surgery was conducted using Exactech GPS navigation (Experimental): The intervention group will include TKA patients whose surgery is conducted with a tibia first gap balancing surgical workflow using the NewtonTM Knee Protocol and navigation-assistance (ExachtechGPS®).
  Interventions: Device: TKA using computer navigation

INTERVENTIONS:
Device: TKA using computer navigation — TKA using Exactech GPS Newton Knee protocol
  Arms: Intervention Group: Patients whose TKA surgery was conducted using Exactech GPS navigation
Procedure: TKA — TKA using manual instrumentation
  Arms: Comparison Group: TKA patients whose surgery was conducted with traditional, manual instrumentation

SUMMARY:
Evaluation of clinical outcomes and patient recovery in patients receiving TKA with traditional instrumentation systems compared to full arc of motion gap balancing using the Newton TM Knee Protocol

DETAILED DESCRIPTION:
The purpose of this study is to evaluate patient outcomes, recovery, and patient/surgeon satisfaction of individuals who undergo a total knee arthroplasty (TKA) using mechanical instrumentation (non-navigated) compared to individuals who undergo a TKA with a tibia first gap balancing surgical workflow using the NewtonTM Knee Protocol and navigation-assistance (ExachtechGPS®).

ELIGIBILITY:
Inclusion Criteria:

* Patients of Kaplan Joint Center, Newton Wellesley Hospital scheduled for TKA with a specific implant

Exclusion Criteria:

* Patients may be excluded due to some medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with TKA using patient reported KOOS JR Questionnaire | Pre-op, 4 weeks post-op, 12 weeks post-op, one year post-op
  The KOOS, JR combines the pain, symptoms, and functional limitations into a single score.
Patient satisfaction with TKA using Oxford Knee Score (OKS) Questionnaire | Pre-op, 4 weeks post-op, 12 weeks post-op, one year post-op
  The OKS is a patient reported questionnaire that measures function and pain with a single score.
Patient satisfaction with TKA using Forgotten Joint Score (FJS) Questionnaire | Pre-op, 4 weeks post-op, 12 weeks post-op, one year post-op
  The Forgotten Joint Score assesses the ability of the patient to forget about their joint given successful treatment by assigning a single score to a series of questions.
Patient recovery from TKA using time from hospital stay to discharge | Post-op measure in hours
  The time of in-patient hospital stay will be measured (in hours).
Patient recovery from TKA by measuring number of outpatient visits | One year post-op
  Number of outpatient visits (scheduled and unscheduled)
Patient recovery from TKA by measuring number of PT visits | One year post-op
  Number of post-op PT visits
Patient recovery from TKA by measuring medication consumption | One year post-op
  Post-op, prescription medication will be recorded in number of pills and dosage
Patient recovery from TKA by measuring use of assisted walking devices | One year post-op
  Patient recovery from TKA by measuring the number of days using an assisted walking device following surgery.

SECONDARY OUTCOMES:
Knee alignment and soft tissue balance | Pre-op, 4 weeks post-op, 12 weeks post-op, one year post-op
  Telemetric x-rays will be used to assess the angles and evaluate the joint line status pre- and post-operatively.
Knee alignment and soft tissue balance | One time (during surgery)
  Patients receiving a TKA NewtonTM Knee, soft-tissue balance will be measured intra-operatively by placing the Newton distractor at the trial reduction stage and acquiring the corresponding joint laxities through the arc of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Joint Center, Newton Wellesley Hospital, Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No